CLINICAL TRIAL: NCT05423015
Title: Elaboration and Assessment of the Effects of Synbiotic on Gut Microbiota Composition of Scholars With Overweight
Brief Title: Assessment of the Effects of Synbiotic on Gut Microbiota Composition in Scholars With Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Diana Patricia Portales-Pérez, Research Professor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 201708
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Childhood Obesity; Childhood Overweight
Keywords: Microbiota; Probiotic; Fermented milk product; Synbiotic
MeSH Terms: conditions — Pediatric Obesity | interventions — Inulin; Fructans

STUDY DESIGN:
Intervention Model Description: Randomised, double blind controlled protocol in children with overweight or obesity aged 6-11 years
Who Masked: Participant, Investigator
Masking Description: The enrolled children were randomized to the three groups in a 1:1:1 ratio stratified by age at the time of study enrolment. The study's investigators and clinical staff were blinded until the final database. Only appointed staff had access to the randomization list to perform labeling of the study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactobacillus casei (Probiotic) (Experimental): Consist in a commercial fermented milk food (Soful LT), which Lactobacillus casei was used as a primary base (probiotic product)
  Interventions: Dietary Supplement: Lactobacillus casei strain Shirota
- L. casei strain Shirota plus inulin (Syn-Inulin) (Experimental): Consist in a commercial fermented milk food (Soful LT), which Lactobacillus casei was used as a primary base (probiotic product) and enriched with 3g of inulin.
  Interventions: Dietary Supplement: Lactobacillus casei strain Shirota plus inulin
- L. casei strain Shirota plus fructans from A. salmiana (Syn-A. salmiana) (Experimental): Consist in a commercial fermented milk food (Soful LT), which Lactobacillus casei was used as a primary base (probiotic product) and enriched with 3g of fructans from A. salmiana.
  Interventions: Dietary Supplement: Lactobacillus casei strain Shirota plus fructans from A. salmiana

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei strain Shirota — Probiotic product were made in a Class II biosafety cabinet. Fifteen milliliters of the fermented milk food wich contains LcS were taken with a sterile syringe, and, at a subsequent time, 15 mL of sterile water were added to the probiotic product.
  Other Names: L. casei Shirota; LcS; Probiotic product
  Arms: Lactobacillus casei (Probiotic)
Dietary Supplement: Lactobacillus casei strain Shirota plus inulin — The Syn-inulin products were made in a Class II biosafety cabinet. Fifteen milliliters of the fermented milk food wich contains LcS were taken with a sterile syringe, and, at a subsequent time, 3 g of inulin (BENEO GmbH) were diluted in 15 mL of sterile water and added to Syn-inulin products.
  Other Names: LcS + inulin; Synbiotic product; Syn-inulin
  Arms: L. casei strain Shirota plus inulin (Syn-Inulin)
Dietary Supplement: Lactobacillus casei strain Shirota plus fructans from A. salmiana — The Syn-A. salmiana products were made in a Class II biosafety cabinet. Fifteen milliliters of the fermented milk food wich contains LcS were taken with a sterile syringe, and, at a subsequent time, 3 g of fructans from A. salmiana were diluted in 15 mL of sterile water and added to Syn-A.salmiana products.
  Other Names: Lactobacillus casei strain Shirota plus A.salmiana; LcS + fructans; LcS + A. salmiana; Synbiotic product; Syn- A. salmiana
  Arms: L. casei strain Shirota plus fructans from A. salmiana (Syn-A. salmiana)

SUMMARY:
This study was a randomized, double-blind controlled protocol in children overweight aged 6-11 years. This study aimed to evaluate the effect of consuming fermented milk products containing Lactobacillus casei strain Shirota (LcS), as a probiotic enriched with prebiotic fructans from A. salmiana or inulin-like standard commercial prebiotic to improve the gut microbiota modulation. After providing detailed information, written informed consent was obtained from parents and written and oral assent from participants before the initial test day. Children were eligible for inclusion in the trial if they were overweight according to the World Health Organization (≥85th body mass index (BMI) percentile for overweight). The trial took place in three full-time elementary schools in San Luis Potosí, México, and the screening of the prospective participants took place up to 1 week prior to the randomization. Children were evaluated over a 6-week intervention period receiving different fermented milk products

DETAILED DESCRIPTION:
Male and female children between the ages of 6- 10 years old were recruited from three schools located in San Luis Potosi, Mexico. According to the World Health Organization, children with overweight were requested to participate and were voluntarily recruited.

After providing detailed information, written informed consent was obtained from parents and written and oral assent from participants before the initial test day. The trial investigated the effect of daily intake of fermented milk products containing Lactobacillus casei strain Shirota (LcS), LcS plus inulin (LcS+inulin), and LcS plus fructans from A. salmiana (LcS+fructans) on gut microbiota composition. The trial protocol was conducted according to the principles of the Declaration of Helsinki. It was approved by the Ethical Committee on Human Experimentation of the State Committee of Health Education and Research of the Health Secretary in San Luis Potosi (register number SLP/012-2017).

ELIGIBILITY:
Inclusion Criteria:

* Children were overweight or obese, according to the World Health Organization (≥85th body mass index (BMI) percentile for overweight, and ≥95th BMI percentile for obesity).

Exclusion Criteria:

* Any known infections, systemic diseases or metabolic diseases, and use of any prescribed medications or antibiotics in the one month before randomization and during the trial.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Gut bacteria associated with changes of the intervention group | Abundance of microbes and relative number of taxa in samples through study completion, 6 weeks intervention of each group
  Comparison of the log2ratio of the genera and the abundance of amplicon sequence variants across the different treatments.
Effect of probiotic and synbiotic products intervention on the BMI z-score | Comparison of BMI-Z score through study completion, 6 weeks intervention of each group.
  Assesment of BMI-Z score changes
Effect of probiotic and synbiotic products intervention on the fat percentage | Comparison of fat percentage through study completion, 6 weeks intervention of each group.
  Assesment of fat percentage changes
Effect of probiotic and synbiotic products intervention on waist and neck circunference | Comparison of waist and neck circunference through study completion, 6 weeks intervention of each group.
  Assesment of waist and neck circunference changes
Effect of probiotic and synbiotic products intervention on glucose, triglycerides and cholesterol serum levels | Comparison of glucose, triglycerides and cholesterol serum levels through study completion, 6 weeks intervention of each group.
  Assesment of glucose, triglycerides and cholesterol serum levels changes

SECONDARY OUTCOMES:
Effect of probiotic and synbiotic products intervention on Free Fatty Acid Receptors (FFAR) 2 and 3 levels | Comparison of mRNA levels of FFAR2 and FFAR3 through study completion, 6 weeks intervention of each group.
  Assessment of mRNA levels of FFAR2 and FFAR3 in the peripheral blood mononuclear cells changes

CONTACTS AND LOCATIONS:
Overall Officials: Diana Patricia Portales-Pérez, phD, Principal Investigator — Universidad Autonoma de San Luis Potosí
Locations (1):
- Facultad de Ciencias Químicas, Universidad Autónoma de San Luis Potosí, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagata S, Asahara T, Ohta T, Yamada T, Kondo S, Bian L, Wang C, Yamashiro Y, Nomoto K. Effect of the continuous intake of probiotic-fermented milk containing Lactobacillus casei strain Shirota on fever in a mass outbreak of norovirus gastroenteritis and the faecal microflora in a health service facility for the aged. Br J Nutr. 2011 Aug;106(4):549-56. doi: 10.1017/S000711451100064X. Epub 2011 Apr 27. PMID 21521545
- [Background] Fernandes R, do Rosario VA, Mocellin MC, Kuntz MGF, Trindade EBSM. Effects of inulin-type fructans, galacto-oligosaccharides and related synbiotics on inflammatory markers in adult patients with overweight or obesity: A systematic review. Clin Nutr. 2017 Oct;36(5):1197-1206. doi: 10.1016/j.clnu.2016.10.003. Epub 2016 Oct 8. PMID 27771020
- [Background] Regalado-Renteria E, Aguirre-Rivera JR, Godinez-Hernandez CI, Garcia-Lopez JC, Oros-Ovalle AC, Martinez-Gutierrez F, Martinez-Martinez M, Ratering S, Schnell S, Ruiz-Cabrera MA, Juarez-Flores BI. Effects of Agave Fructans, Inulin, and Starch on Metabolic Syndrome Aspects in Healthy Wistar Rats. ACS Omega. 2020 May 6;5(19):10740-10749. doi: 10.1021/acsomega.0c00272. eCollection 2020 May 19. PMID 32455193
- [Background] Larsen N, Vogensen FK, Gobel RJ, Michaelsen KF, Forssten SD, Lahtinen SJ, Jakobsen M. Effect of Lactobacillus salivarius Ls-33 on fecal microbiota in obese adolescents. Clin Nutr. 2013 Dec;32(6):935-40. doi: 10.1016/j.clnu.2013.02.007. Epub 2013 Mar 4. PMID 23510724
- [Background] Martinez-Gutierrez, F., Ratering, S., Juárez-Flores, B., et al. Potential use of Agave salmiana as a prebiotic that stimulates the growth of probiotic bacteria. Lwt, 2017; 84:151-159.
- [Background] Nagata S, Chiba Y, Wang C, Yamashiro Y. The effects of the Lactobacillus casei strain on obesity in children: a pilot study. Benef Microbes. 2017 Aug 24;8(4):535-543. doi: 10.3920/BM2016.0170. Epub 2017 Jun 16. PMID 28618860
- [Background] Safavi M, Farajian S, Kelishadi R, Mirlohi M, Hashemipour M. The effects of synbiotic supplementation on some cardio-metabolic risk factors in overweight and obese children: a randomized triple-masked controlled trial. Int J Food Sci Nutr. 2013 Sep;64(6):687-93. doi: 10.3109/09637486.2013.775224. Epub 2013 Mar 12. PMID 23477506
- [Derived] Vega-Cardenas M, Martinez-Gutierrez F, Lara-Ramirez EE, Reynaga-Hernandez E, Yanez-Estrada L, Ratering S, Schnell S, Godinez-Hernandez CI, Vargas-Morales JM, Portales-Perez DP. Agave fructans enhance the effects of fermented milk products on obesity biomarkers: a randomised trial. Benef Microbes. 2023 Apr 18;14(2):153-164. doi: 10.3920/BM2022.0078. Epub 2023 Mar 1. PMID 36856122